CLINICAL TRIAL: NCT05419934
Title: Is Eye-Movement Desensitization and Reprocessing (EMDR) Therapy Effective in Children Aged 3 to 6 Years With Trauma-related Disorders or Stressors and Anxiety? A Double-blinded Randomized Controlled Trial.
Brief Title: EMDR Therapy in Young Children, a Double-blinded Randomized Controlled Trial
Acronym: EMDRJEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-HPNCL-09
Record Dates: First submitted 2022-06-02; First posted 2022-06-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Trauma, Psychological; Stress, Psychological; Anxiety Disorders
MeSH Terms: conditions — Psychological Trauma; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMDR (Experimental): Patient receiving " EMDR therapy " over 6 to 12 sessions.
  Interventions: Behavioral: EMDR therapy
- CBT Control Therapy (Sham Comparator): Patient receiving the " CBT Control Therapy " over 6 to 12 sessions
  Interventions: Behavioral: CBT Control therapy

INTERVENTIONS:
Behavioral: EMDR therapy — Children will receive an EMDR psychotherapy comprising 8 treatment phases. As the treatment progresses, the child will proceed to desensitize the events of adversity experienced.
  Phase 1 and 2, before the desensitization phases:
  1. History of the patient (collection of anamnesis)
  2. Securing the patient, preparing for the desensitization phases
     Desensitization phases, to be repeated for each traumatic event to be desensitized:
  3. Evaluation of the target to be treated
  4. Desensitization
  5. Installation of positive beliefs
  6. Body scanner (verification of body non-response)
  7. Closure, verification that the patient is in a stable emotional state allowing him to leave the session
     Reassessment phase, to be repeated for each traumatic event that has been desensitized:
  8. Reassessment of the traumatic target, verification of complete desensitization.
  Arms: EMDR
Behavioral: CBT Control therapy — Children in the control group receive Cognitive Behavioral Therapy (CBT) administered by the Lenval Foundation (CHU de Nice - France) within the Pediatric Psychotrauma Assessment Center (Centre d'évaluation du psychotraumatisme pédiatrique - CE2P).Cognitive and behavioral therapies are a standard treatment in the care service. Children in the control group will receive CBT specific to the treatment of PTSD in children under 6 years of age. CBT treatments dedicated to early childhood trauma have already been tested in the United States, and have shown evidence of effectiveness in randomized controlled trials (Mc Guire et al., 2021; Scheeringa et al., 2011).
  Arms: CBT Control Therapy

SUMMARY:
This project aims to answer to the question of EMDR effectiveness in young children and to determine whether or not the therapy effectiveness is related to the level of cognitive functioning in young children. The study requires a total of 60 children, girls and boys, aged 3 to 6 years and presenting disorders related to stressors, anxiety and/or trauma. Participants will be randomly distributed in two groups: "EMDR therapy" (N=30) group or "control therapy" (N=30) group. The study will take place in four stages: 1/ Pre-treatment phase : An evaluation of child's various cognitive and executive functions, child's symptomatology and parental distress is planned in a pre-treatment phase. 2/ Treatment phase : An EMDR therapy or a routine care is administered to the child between 6 to 10 weeks. 3/ Post-treatment phase : A reassessment of child's and parent's symptoms is planned at the end of treatment. 4/ Continuation of treatment: Children who have received control therapy and without symptomatic improvement will be proposed EMDR treatment. These children will receive the same symptomatic assessments at the end of EMDR treatment.

A significant reduction in disorders related to trauma or stress and anxiety factors and their symptomatology, as well as comorbid disorders and their symptomatology, is expected in children who received EMDR therapy compared to the group who received a control therapy. These results are expected to be robust over a period of at least 3 months. The positive effects of EMDR on child symptomatology are also expected to be more pronounced in children showing higher levels of cognitive functioning

DETAILED DESCRIPTION:
Eye-Movement Desensitization and Reprocessing (EMDR) therapy is now recommended to anyone suffering from emotional disturbance related to psychological trauma, including babies and very young children. Results of this therapy are promising in young children for PTSD and its comorbidities. However, no studies have documented yet the specific effects of individual EMDR therapy in the 3-6 years children.

The question of the EMDR effectiveness in this population should be investigated first to meet the therapeutic needs in the care management of childhood psychotrauma, and secondly because EMDR therapy involves memory and executive functions that are very immature in children under 6 years old.

Indeed, EMDR involves therapeutic methods such as cognitive restructuring which requires that certain executive functioning components to be functional, even those processes are still developing in young children. EMDR also involves an exposure in the imagination that solicits episodic memories, whereas the ability of young children to retrieve thoses memories is very limited compared to that of adults. Finally, the alternating bilateral stimuli used in EMDR would have an effect on autobiographical memory. However, an infantile amnesia is observed between the ages of 2 and 6, with an absence and then a poverty of autobiographical memories.

Therefore, the present project aims to answer to the question of EMDR effectiveness in young children suffering from stress related disorders, anxiety and/or trauma, but also to determine whether or not the therapy effectiveness is related to the level of cognitive functioning in young children. This study requires a total of 60 children, girls and boys, aged 3 to 6 years and presenting disorders related to stressors, anxiety and/or trauma. Participants will be randomly distributed in two groups: "EMDR therapy" (N=30) group or "control therapy" (N=30) group. The study will take place in four stages: 1/ Pre-treatment phase : An evaluation of child's various cognitive and executive functions, child's symptomatology and parental distress is planned in a pre-treatment phase. 2/ Treatment phase : An EMDR therapy or a routine care is administered to the child between 6 to 10 weeks. 3/ Post-treatment phase : A reassessment of child's and parent's symptoms is planned at the end of treatment. 4/ Continuation of treatment: Children who have received control treatment and without symptomatic improvement will be proposed EMDR treatment. These children will receive the same symptomatic assessments at the end of EMDR treatment.

In terms of results, a significant reduction in disorders related to trauma or stress and anxiety factors and their symptomatology, as well as comorbid disorders and their symptomatology, is expected in children who received EMDR therapy compared to the group who received a control therapy. These results are expected to be robust over a period of at least 3 months. The positive effects of EMDR on child symptomatology are also expected to be more pronounced in children showing higher levels of cognitive functioning.

This protocol represents the first randomized controlled trial to investigate effects of an individual EMDR therapy conducted specifically in children aged 3 to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3 to 6 at the time of inclusion;
* Established diagnosis of one or more disorders related to a trauma or a stress factor, and/or an anxiety disorder, assessed by the Diagnostic Infant and Preschool Assessment (DIPA) diagnostic tool
* Typical language

Exclusion Criteria:

* Child taking a psychotropic treatment
* Suicidal intentions or ideation of the main caregivers, or of the child, and self-harming behavior;
* Parent(s) or care figure(s) with a substance use disorder;
* Presence or diagnosis of specific pathological conditions in the child (neurodevelopmental disorders based on Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria, brain trauma, or neurological pathology);
* Participation of the child in another biomedical research on the psychic care of disorders related to trauma or stress and anxiety factors

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Diagnostic Infant and Preschool Assessment at 3months | at 3 months from inclusion
  diagnostic of 13 pathologies, such as post Traumatic stress disorder (PTSD) or others stress related disorders, Anxiety related disorders, and associated disorders. This tool as 517 items. This scale doesn't work on numerical values (there is no min, max or cut scores), this scale makes it possible to confirm or invalidate the presence of symptoms necessary for establishing diagnoses on Diagnosis and Statistical Manual of Mental Disorders (DSMV) criteria.
Diagnostic Infant and Preschool Assessment at 6 months | at 6 months from inclusion
  diagnostic of 13 pathologies, such as post Traumatic stress disorder (PTSD) or others stress related disorders, Anxiety related disorders, and associated disorders. This tool as 517 items. This scale doesn't work on numerical values (there is no min, max or cut scores), this scale makes it possible to confirm or invalidate the presence of symptoms necessary for establishing diagnoses on Diagnosis and Statistical Manual of Mental Disorders (DSMV) criteria.

SECONDARY OUTCOMES:
Preschool Anxiety Assessment | at inclusion, at 3 and 6 months from inclusion
  symptoms of anxiety is measure by Preschool Anxiety Scale (PAS) The PAS is a heteroevaluation (for parents or the main care figure) to assess symptomatology of anxiety in children aged 3 to 6 years. This tool has 34 items, based on a 5-points Likert scale, each item is scored from 0 to 4, the PAS has a score ranging from 0 to 112. To interpret this questionnaire, T-scores must be used. T-Scores enable the comparison of a child scores against norms from an equivalent age and gender group from a representative normative sample.
Parental Stress | at inclusion, at 3 and 6 months from inclusion
  symptoms of parental distress and parent-child dysfunctional interaction is performed by Parental Stress Index Screening Form (PSI-SF). The "Parental Stress Index Short Form" is a self-assessment intended for the child's parent The PSI-SF has 36 items from the original 120-item PSI and based on a 5-points Likert scale, each item is scored from 1 to 5, the PSI-SF has a score ranging from 36 to 180. Percentile scores are used to interpret the scores.
  Scores at or above the 85th percentile are considered high (normal range : 15th-80th percentile)
symptoms of Post Traumatic Stress Disorder | at inclusion, at 3 and 6 months from inclusion
  measure of symptoms of PTSD by Young Child Post-traumatic Stress Disorder Checklist.
  This scale aims to screen for post-traumatic stress disorder symptoms in children aged 1 to 6 years old, by evaluating traumatic exposures (13 items), symptoms presented by the child (23 items) and his level of impairment or functional impairment (6 items). Items 14 to 36 relate to symptoms of PTSD and are based on a 5-points Likert scale, each item is scored from 0 to 4, the YCPC has a score ranging from 0 to 92. The diagnosis Cutoff is at 26 or more for items 14-36, it indicates a "probable diagnosis" of PTSD. Items 37 to 42 study functional impairment. These items scores can be added together to form a disability score, but they are not used in the PTSD symptom score
Child Behavior | at inclusion, at 3 and 6 months from inclusion
  pathologic behaviors are measured by Child Behavior Checklist " (CBCL) ;
  The Child Behavior Checklist assesses anxiety, depression, emotional dysregulation, sleep disorders, attention problems, withdrawal behavior, and aggressive behavior. This list of items initially used with children aged 6 to 18 has been adapted for preschoolers. The study plans to use the preschool form (CBCL/ 1.5-5) for children aged 3 years to 5 years and 11 months, and the original CBCL for children aged 6 years to 6 years and 11 months.
  The Checklist is based on a 3-points Likert scale, each item is scored from 0 to 2, the CBCL has a score ranging from 0 to 230.
  To interpret this questionnaire, T-scores must be used.
cognitive function | at inclusion
  use of French version of the Wechsler Preschool and Primary Scale of Intelligence ; only the subtests: Picture naming - for children ages 3 to 6 years ; Matrix - for children ages 4 to 6 years; Pictures Memory - for children ages 3 to 3 years and 11 months; Spatial Memory (Zoo location)- for children ages 3 to 6 years;
  The Wechsler Preschool and Primary Scale of Intelligence (WPPSI) is a cognitive assessment of children aged 2 years and 6 months to 7 years and 7 months. The 4th revision makes it possible to take into account the major stages of the child's cognitive and neurological development. Only subtests that show how the child develops certain major cognitive functions will be administered
executive functioning | at inclusion
  cognitive functioning (executive functioning) measure by french test of Executive Function Assessment Battery for Preschoolers named " La batterie d'évaluation des fonctions exécutives pour enfants d'âge préscolaire " (BEFEX-P) version 4.0 - (Monette & Bigras, 2017)
  This evaluation includes two independent tests: a Stroop test adapted to the child, and a tracing tracks. The Stroop fruit is an evaluation of inhibition and flexibility functions in preschool children which is practiced in verbal condition.
  Trace tracing is a cognitive task that allow the evaluation of executive functions (inhibition and flexibility) in preschool children.
autobiographical memory | at inclusion
  cognitive functioning (autobiographical memory) measure with french test of Autobiographical Memory Evaluation Task named " Tâche d'Evaluation de la Mémoire Autobiographique " (TEMA ; Deplus, de Romree, & Van Broeck, 2013)
  The TEMA assessment evaluates the functioning of autobiographical memory in preschool children (children from 3 years to 5 years and 11 months). This test makes the child do exercises to produce autobiographical memories.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France